CLINICAL TRIAL: NCT06055374
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Efficacy of BxC-I17e Administered Subcutaneously in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Investigate the Safety, Tolerability, and Efficacy of BxC-I17e Repeated-dose SC Injection in Patients With Moderate to Severe Atopic Dermatitis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was integrated into BRE-AD01-001 study
Sponsor: Brexogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BRE-AD01-002
Record Dates: First submitted 2023-09-12; First posted 2023-09-26 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BxC-I17e (Experimental): * Subcutaneous (SC) injection of 50, or 100 ug BxC-I17e
  * Treatment on Day 1, 15, 29, and 43 for a total 4 biweekly doses
  Interventions: Drug: BxC-I17e
- Placebo (Placebo Comparator): * Subcutaneous (SC) injection of the matching placebo
  * Treatment on Day 1, 15, 29, and 43 for a total 4 biweekly doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BxC-I17e — Pharmaceutical form : solution for injection
  Arms: BxC-I17e
Drug: Placebo — Pharmaceutical form : solution for injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and efficacy of a multiple SC dose of BxC-I17e in patients with moderate to severe atopic dermatitis (AD)

ELIGIBILITY:
Inclusion Criteria:

1. Patients (males or females) aged 18 years or older
2. Patients have documented history of moderate to severe AD, that has been present for at least 1 year
3. History of inadequate response to a stable regimen of TCSs or TCIs as treatment for AD
4. Patients must agree to apply stable doses of additive-free, basic bland emollient lotions twice daily for at least 7 days before the Baseline Visit
5. Willingness and ability to comply with clinic visits and study-related procedures
6. Patients should be able to read, understand, and be willing to sign the ICF

Exclusion Criteria:

1. Presence of any of the following laboratory abnormalities

   * Hemoglobin < 11 g/dL
   * WBC < 3.5 × 103/μL
   * Platelet count < 125 × 103/μL
   * Neutrophils < 1.75 × 103/μL
   * AST/ALT > 1.5 × ULN
   * Total bilirubin > ULN
   * Creatinine > ULN
   * Creatine phosphokinase > ULN
2. Positive test for hepatitis B surface antigen, and/or hepatitis C antibody
3. Active dermatologic conditions that may confound the diagnosis of AD
4. Prior exposure to any investigational systemic treatment or is currently enrolled in another clinical study
5. Significant concomitant illness or history of significant illness such as cardiac, renal, neurological, endocrinological, metabolic or lymphatic disease, or any other illness or condition that would adversely affect the patient's participation in this study
6. Treatment with TCS, and/or TCI, within 1 week prior to the Baseline Visit
7. Known history of human immunodeficiency virus (HIV) infection
8. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Baseline to Week 26
  Incidence of treatment-emergent adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Incidence, severity and relationship of adverse events(AEs) | Baseline to Week 26
  Incidence, severity and relationship of adverse events as assessed by CTCAE v5.0
Number of abnormalities and change from baseline in Vital signs | Baseline to Week 26
  Supine blood pressure and pulse rate, tympanic temperature, and respiratory rate
Number of abnormalities in 12-lead electrocardiogram (ECG) | Baseline to Week 26
  PR interval, QRS interval, RR interval, QT interval and QT interval using Friderica's correction (QTcF)
Number of abnormalities in clinical laboratory parameter | Baseline to Week 26
  Hematology, clinical chemistry, and urinalysis parameters
Frequency and proportion of clinically significant finding of physical examination | Baseline to Week 26
  Assessments of the following body categories : skin, HEENT (head, eye, ears, nose, and throat), cardiovascular, respiratory, gastrointestinal, endocrine/metabolic, genitourinary, psychiatric, hematologic/lymphatics, musculoskeletal, neurologic, hepatic, and allergic/immunologic
Proportion of patients who achieved the Investigator's Global Assessment (IGA) score of 0 or 1 | Baseline to Week 14
  The IGA is an assessment instrument used in clinical studies to rate the severity of Atopic dermatitis globally, based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Change and percent change in Body Surface Area (BSA) | Baseline to Week 14
  The BSA affected by atopic dermatitis will be assessed for each major section of the body (head, trunk, arms, and legs). Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
Change and percent change in Eczema Area and Severity Index (EASI) | Baseline to Week 14
  The EASI is a composite index with scores ranging from 0 to 72. Higher scores indicates worse condition.
Change and percent change in Scoring Atopic Dermatitis (SCORAD) | Baseline to Week 14
  The SCORAD is a clinical tool for assessing the severity of Atopic dermatitis. Total score ranged from 0 (absent disease) to 103 (severe disease).
Change and percent change in Pruritus Numerical Rating Scale (NRS) | Baseline to Week 14
  The Pruritus NRS is a simple assessment tool used to report the intensity of their pruritus (itch) ranges from 0 to 10 with 0 being 'no itch' and 10 being the' worst itch imaginable.
Change and percent change in Dermatology Life Quality Index (DLQI) | Baseline to Week 14
  The DLQI is a validated questionnaire designed to measure the impact of skin disease on the Quality of Life. The higher the score, the greater the impact is on the quality of life
Change and percent change in Patient-Oriented Eczema Measure (POEM) | Baseline to Week 14
  The POEM is a validated 7-item questionnaire used to assess disease symptoms with a scoring system of 1 to 28. The higher score, the higher morbidity.
Changes in the level of eosinophils in the serum and correlation with other parameters | Baseline to Week 14
  The level of biomarkers in serum
Changes in the level of Thymus Activation Regulated Chemokine (TARC) in the serum and correlation with other parameters | Baseline to Week 14
  The level of biomarkers in serum
Changes in the level of Pulmonary Activation-Regulated Chemokine (PARC) in the serum and correlation with other parameters | Baseline to Week 14
  The level of biomarkers in serum
Changes in the level of eotaxin-3 in the serum and correlation with other parameters | Baseline to Week 14
  The level of biomarkers in serum
Changes in the level of Macrophage-Derived Chemokine (MDC) in the serum and correlation with other parameters | Baseline to Week 14
  The level of biomarkers in serum
Changes in the level of periostin in the serum and correlation with other parameters | Baseline to Week 14
  The level of biomarkers in serum
Changes in the level of total Immunoglobulin E (IgE) in the serum and correlation with other parameters | Baseline to Week 14
  The level of biomarkers in serum
Changes in the level of total Interleukin-13 (IL-13) in the serum and correlation with other parameters | Baseline to Week 14
  The level of biomarkers in serum
Changes in the level of total Interleukin-22 (IL-22) in the serum and correlation with other parameters | Baseline to Week 14
  The level of biomarkers in serum
Changes in the level of total Interleukin-31 (IL-31) in the serum and correlation with other parameters | Baseline to Week 14
  The level of biomarkers in serum

IPD SHARING:
Plan to Share IPD: No